CLINICAL TRIAL: NCT04491461
Title: Acute Effects of an Herbal Tea Blend on Immune Surveillance and Activation Status of Natural Killer Cells.
Brief Title: Acute Effects of an Herbal Tea on Immune Surveillance and Activation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 152-018
Record Dates: First submitted 2020-07-26; First posted 2020-07-29 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-06

CONDITIONS: Active Immune Response

STUDY DESIGN:
Intervention Model Description: The study uses a randomized double-blinded controlled cross-over study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herbal tea blend (Active Comparator): 1 cup of herbal tea blend containing Rosehip and other berry extracts.
  Interventions: Dietary Supplement: Herbal tea blend
- Warm water (Sham Comparator): 1 cup of warm water.
  Interventions: Dietary Supplement: Warm water

INTERVENTIONS:
Dietary Supplement: Herbal tea blend — 1 cup of freshly brewed tea from an herbal tea blend.
  Arms: Herbal tea blend
Dietary Supplement: Warm water — 1 cup of warm water
  Arms: Warm water

SUMMARY:
A small cross-over trial on 24 people involving an herbal tea blend to test whether consuming 1 cup of tea triggers changes in the numbers of natural killer cells in the blood circulation as evidence of immune cell trafficking within 2 hours.

DETAILED DESCRIPTION:
A randomized, cross-over, controlled study design will be used to evaluate the effects of consumption of 1 cup of an herbal tea blend to consumption of the same volume of warm water. The study is of 3 weeks' duration, with evaluation of the herbal tea blend versus warm water at week 1 and week 2 with a one week washout between visits. On each visit, a baseline blood draw is performed, followed by consuming of the herbal tea blend or warm water. Blood draws are performed at 1 and 2 hours after consumption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults;
* Age 18-75 years (inclusive);
* Veins easy to see in both arms (to allow for the multiple blood draws);
* Willing to comply with a 24-hour wash-out period for vitamins and nutritional supplements;

Exclusion Criteria:

* Previous major gastrointestinal surgery (absorption of test product may be altered) (minor surgery not a problem, including previous removal of appendix and gall bladder);
* Taking anti-inflammatory medications on a daily basis;
* Currently experiencing intense stressful events/ life changes;
* Currently in intensive athletic training (such as marathon runners);
* Currently taking antipsychotic medications such as clozapine, Risperdal, Abilify, Zyprexa or Seroquel;
* Actively depressed;
* An unusual sleep routine (examples: working graveyard shift, irregular routine with frequent late nights, studying, partying);
* Unwilling to maintain a constant intake of supplements over the duration of the study;
* Anxiety about having blood drawn;
* Women of childbearing potential: Pregnant, nursing, or trying to become pregnant;
* Known food allergies related to ingredients in active test product.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-12-19 (Actual)

PRIMARY OUTCOMES:
Change to natural killer cell numbers in blood circulation | Changes at 1 and 2 hours after consumption
  Flow cytometry evaluation of natural killer cell numbers

SECONDARY OUTCOMES:
Change to natural killer cell activation status | Changes at 1 and 2 hours after consumption
  Flow cytometry evaluation of CD69 expression on natural killer cells in the blood circulation

CONTACTS AND LOCATIONS:
Overall Officials: GITTE JENSEN, Study Director — NIS Labs
Locations (1):
- Gitte Jensen, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No